CLINICAL TRIAL: NCT00196482
Title: Impact of Human Milk Fortifiers on Acid-Base Status in Preterm Infants
Brief Title: Human Milk Fortifiers and Acid-Base Status
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Collaborators: NUMICO,Dr. Heike Mueller, Friedrichsdorf, Germany (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Fortifier 01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2006-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Premature Birth
Keywords: growth; oral feeding; nutrition
MeSH Terms: conditions — Premature Birth

INTERVENTIONS:
Drug: changing of fortifier

SUMMARY:
Double-blind randomized controlled trial to investigate the impact of two human milk fortifiers on acid-base status and longitudinal growth and weight gain in preterm infants.

Two different compositions are tested, main difference is in electrolyte composiiton.

DETAILED DESCRIPTION:
Two groups each consisting of 15 infants with a birth weight below 2000g are studied.randomization is startified by three birth weigth classes (<1000g, 1000-1500g,1500 - 2000g) human milk fortifier is introduced in two steps after oral feeding is achieved. two acid-base status and electrolyte concentrations are measured. when metabolic acidosis, defined as BE < -6 mmol/l, occurs fortifier feeding is stopped, and after a wash-out period of three days the alternative product is used.again, occurence of metabolic acidosis, need for oral bicarbonate and effect on longitudinal growth an weight gain are registered.

ELIGIBILITY:
Inclusion Criteria:

growing premature infants with a birth weight < 2000g

Exclusion Criteria:

congenital malformation chromosomal disorders sepsis metabolic disorders need for mechanical ventilation

Ages: 10 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30
Dates: Start 2004-06; Study Completion 2006-02

PRIMARY OUTCOMES:
frequency of metabolic acidosis

SECONDARY OUTCOMES:
need for oral bicarbonate administartion
longitudinal growth
weight gain
amino acid levels in plasma an urine

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Fusch, Study Chair — Department of Neonatology, University Hospital Greifswald
Locations (1):
- University Hospital, Greifswald, M-V, Germany

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765